CLINICAL TRIAL: NCT02751359
Title: Characterization of the Analgesic Effects of Oral CBD in Healthy, Normal Volunteers
Brief Title: Characterization of the Analgesic Effect of CBD in Healthy, Normal Volunteers
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: INSYS Therapeutics Inc (Industry)
Responsible Party: Principal Investigator, Ziva D. Cooper, PhD, Associate Professor of Clinical Neurobiology (in Psychiatry), University of California, Los Angeles
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: 7009
Record Dates: First submitted 2016-04-12; First posted 2016-04-26 (Estimated); Results first posted 2021-05-12 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — Cannabidiol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active CBD (Active Comparator): Each subject will receive each active dose of cannabidiol, one active dose per 3 of the 4 study days. The active cannabidiol doses include 200, 400 and 800 mg of cannabidiol.
  Interventions: Drug: Cannabidiol
- Placebo (Placebo Comparator): On 1 of the 4 study days, participants will receive placebo cannabidiol (0 mg)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cannabidiol — 200, 400, or 800 mg Cannabidiol
  Other Names: CBD
  Arms: Active CBD
Drug: Placebo — 0 mg Cannabidiol
  Arms: Placebo

SUMMARY:
The purpose of this double-blind, placebo-controlled study is to determine the analgesic effects of cannabidiol (CBD), a chemical constituent found in cannabis that does not have intoxicating effects. The analgesic effects of CBD will be assessed using the Cold-Pressor Test (CPT), a laboratory model of pain which has predictive validity for the clinical use of analgesics.

DETAILED DESCRIPTION:
This within-subject, double-blind, placebo-controlled study will assess the analgesic and subjective effects of a range of CBD doses (0, 200, 400, or 800 mg, po). Volunteers will participate in 4 outpatient laboratory sessions over the course of 4 weeks during which the analgesic effects of CBD will be assessed using the Cold-Pressor Test (CPT), a laboratory model of pain which has predictive validity for the clinical use of analgesics. The order of CBD dose will be randomized across participants. Secondary measures will include subjective and physiologic effects of CBD.

ELIGIBILITY:
Inclusion Criteria:

* Able to perform study procedures
* Women practicing an effective form of birth control

Exclusion Criteria:

* Female subjects who are currently pregnant or breastfeeding.
* Current illicit drug use
* Presence of significant medical illness
* History of heart disease
* Request for drug treatment
* Current parole or probation
* Recent history of significant violent behavior
* Major psychiatric disorder
* Current use of any prescription or over-the-counter medication
* Current pain
* Clinically significant Raynaud's syndrome

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2020-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ziva D Cooper, PhD, Principal Investigator — New York State Psychiatric Institute / CUMC
Locations (1):
- Cooper, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Group - Repeated Measures: Each subject will receive each active dose of cannabidiol, one active dose per 3 of the 4 study day; on 1 of the 4 study days, participants will receive placebo cannabidiol (0 mg).
Period: Overall Study
Arm/Group | Single Group - Repeated Measures
Started | 18
Completed | 17
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Demographics were collected for study completers
Arm/Group | Single Group - Repeated Measures
Number analyzed (Participants) | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 2
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Analgesia: Change From Baseline in Pain Tolerance and Threshold as Measured by the Cold Pressor Test
Description: Time to first feel pain ("Pain threshold" measured in seconds) during the Cold Pressor Test and withdraw the hand from the cold water ("Pain Tolerance" measured in seconds). Changes in threshold from baseline were averaged across study sessions for each CBD dose.
Time Frame: Baseline, 60 minutes, 120 minutes 180 minutes, 240 minutes, 300 minutes and 360 minutes after each dose
Measure: Mean (Standard Error); unit: Seconds
Groups:
- Active CBD 200 mg: Cannabidiol: 200mg
- Active CBD 400 mg: Cannabidiol: 400mg
- Active CBD 800 mg: Cannabidiol: 800mg
Arm/Group | Active CBD 200 mg | Active CBD 400 mg | Active CBD 800 mg | Placebo
Number analyzed (Participants) | 17 | 17 | 17 | 17
Seconds
  Threshold | 9.7 (7.0) | 2.2 (0.8) | 2.1 (2.4) | 1.2 (0.9)
  Tolerance | 5.1 (5.3) | 15.3 (8.0) | -0.6 (0.9) | 9.6 (5.3)

2. Secondary Outcome: Subjective Drug Effects Related to Abuse Liability as Measured by Visual Analog Scales
Description: Participants rate the strength of their desire to take again, drug liking, good effect and bad effect. Each item was presented and the participant was asked to rate his / her rating on a scale anchored by 'Not At All' (0 mm) to 'Extremely' (100 mm). The average of all timepoints is reported for each category.
Time Frame: 30 minutes, 60 minutes, 90 minutes, 120 minutes, 150 minutes, 180 minutes, 210 minutes, 270 minutes, 300 minutes, 330 minutes, 360 minutes
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active CBD 200 mg | Active CBD 400 mg | Active CBD 800 mg | Placebo
Number analyzed (Participants) | 17 | 17 | 17 | 17
score on a scale
  Good effect | 8.7 (3.8) | 19.0 (5.9) | 10.2 (4.7) | 13.3 (5.7)
  Bad effect | 5.7 (3.5) | 9.1 (4.4) | 4.5 (2.2) | 4.1 (2.5)
  Drug liking | 18.7 (5.2) | 21.3 (5.7) | 15.8 (5.1) | 18.8 (6.1)
  Desire to take again | 17.9 (5.7) | 23.6 (6.6) | 18.1 (5.9) | 17.5 (6.1)

ADVERSE EVENTS:
Time Frame: During and after each study session, average of 4 weeks total study participation
Arm/Group | Active CBD 200 mg | Active CBD 400 mg | Active CBD 800 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/17 | 0/18
Other Adverse Events (participants affected / at risk) | 5/18 | 10/18 | 7/17 | 7/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active CBD 200 mg (N=18) | Active CBD 400 mg (N=18) | Active CBD 800 mg (N=17) | Placebo (N=18)
Lethargy (General disorders) | 5 | 5 | 5 | 5
Gas and cramps (Gastrointestinal disorders) | 1 | 4 | 4 | 1
Subtle mood change (General disorders) | 0 | 0 | 0 | 1
Frequent urination (Renal and urinary disorders) | 0 | 1 | 0 | 0
Wooziness (General disorders) | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-23): https://cdn.clinicaltrials.gov/large-docs/59/NCT02751359/Prot_SAP_000.pdf